CLINICAL TRIAL: NCT04844372
Title: Impact of Regional Anesthesia on Blood Pressure in Lower Limb Traumatism : IRB (Impact of Regional Anesthesia on Blood Pressure)
Brief Title: Impact of Regional Anesthesia on Blood Pressure in Lower Limb Traumatism
Acronym: IRB
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0091
Record Dates: First submitted 2021-04-06; First posted 2021-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Fracture, Ankle; Fracture Leg
Keywords: Surgery for Ankle and/or leg fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the hemodynamic impact of two anaesthetic strategies 'Regional anesthesia' versus 'General anesthesia' in leg and ankle fractures surgery.

DETAILED DESCRIPTION:
Leg and/or ankle surgery is frequently performed under General Anesthesia (GA). GA is frequently associated with a high risk of hypotension with significant consequences.

Regional anesthesia could be an interesting alternative to GA in order to limit hemodynamic consequences, especially in elderly patients.

Furthermore, in the current state of Covid 19 crisis, regional anesthesia could provide solutions in preserving drugs for GA and exposing less medical staff on patient's airway.

Currently, unlike neuraxial anesthesia, few data deal with impact of peripheral RA and hemodynamic consequences.

The investigators hypothesize that the use of Regional anesthesia reduces the use of intraoperative vasopressor.

After ethical committee approval, a retrospective cohort of patients with lower limb traumatism, in Montpellier's University Hospital, was analyzed from 2016 to 2020. An informational note was given to all patients participating to the study.

ELIGIBILITY:
Inclusion criteria

* ASA I - IV
* Ankle and/or leg fracture
* Operated between january 2016 and december 2020 at Montpellier

Exclusion criteria

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Surgical revision or surgery for pre-existing infection, tumour
  * Intubated patient / unconscious patient
  * Vasopressors before surgery
  * Haemostasis disorder
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
use of vasopressors | during surgery
  use of vasopressors during surgery

SECONDARY OUTCOMES:
Total dose of vasoconstrictor | during surgery
  Total dose of vasoconstrictor administered
Duration of peroperative hypotension | during surgery
  Duration of peroperative hypotension
Post-operative complications | up to 7 days
  Nausea/vomiting ; Cardiovascular complications ( dysrhythmias, ischaemia, Complications related to regional anesthesia (sciatic nerve paralysis, femoral) haematoma thromboembolism, sepsis, postoperative cognitive disorders);

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas SURCIN-TSEKOURAS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC